CLINICAL TRIAL: NCT01262560
Title: Phase II Randomized Trial of Prophylactic Manuka Honey for the Reduction of Chemoradiation Therapy Induced Esophagitis-Related Pain During the Treatment of Lung Cancer
Brief Title: Manuka Honey in Preventing Esophagitis-Related Pain in Patients Receiving Chemotherapy and Radiation Therapy For Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RTOG 1012; RTOG-1012; CDR0000690182; NCI-2011-02620 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Dysphagia; Lung Cancer; Pain; Esophagitis
Keywords: pain; dysphagia; recurrent non-small cell lung cancer; stage IA non-small cell lung cancer; stage IB non-small cell lung cancer; stage IIA non-small cell lung cancer; stage IIB non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent small cell lung cancer; esophagitis
MeSH Terms: conditions — Deglutition Disorders; Lung Neoplasms; Pain; Esophagitis; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Supportive Care (Active Comparator): Standard supportive care
  Interventions: Drug: Standard supportive care
- Liquid Manuka Honey (Experimental): Manuka honey in liquid form
  Interventions: Drug: Manuka honey in liquid form
- Lozenge Manuka Honey (Experimental): Manuka honey in lozenge form
  Interventions: Drug: Manuka honey in lozenge form

INTERVENTIONS:
Drug: Manuka honey in liquid form — Patients swallow 10 cc (approximately 2 level teaspoons) of liquid Manuka honey 4 times per day while awake over an approximately 12 hour period (e.g. 8 a.m., Noon, 4 p.m., and 8 p.m.) 7 days/week during concurrent chemotherapy and radiation treatment.
  Arms: Liquid Manuka Honey
Drug: Manuka honey in lozenge form — Patients place 2 lozenges (the equivalent of 10 cc of liquid Manuka honey), one at a time, in the mouth, allowing each lozenge to dissolve on the tongue/in the mouth, swallowing the honey as it dissolves. Patients do this 4 times per day while awake over an approximately 12 hour period (e.g. 8 a.m., Noon, 4 p.m., and 8 p.m.) 7 days/week during concurrent chemotherapy and radiation treatment.
  Arms: Lozenge Manuka Honey
Drug: Standard supportive care — Patients receive standard supporting care for esophagitis-related pain as needed during concurrent chemotherapy and radiation treatment. The following regimen is recommended, but the local standard of care is permitted.
  1. A compound containing viscous lidocaine and magnesium aluminum oxide (Maalox®);
  2. Liquid or solid oxycodone, 5-10 mg, every 3 hours as needed.
  Arms: Supportive Care

SUMMARY:
RATIONALE: Manuka honey may prevent or reduce esophagitis-related pain caused by chemotherapy and radiation therapy. It is not yet known whether Manuka honey is more effective than standard care in preventing pain.

PURPOSE: This randomized phase II clinical trial is studying Manuka honey to see how well it works in preventing esophagitis-related pain in patients receiving chemotherapy and radiation therapy for lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the relative efficacy of 4 times a day consumption of liquid or lozenge Manuka honey to delay or prevent radiation esophagitis-related pain (during combined chemotherapy and radiation therapy for lung cancer) as compared to standard supportive treatment, as measured at week 4 by Numerical Rating Pain Scale (NRPS) for pain upon swallowing.

Secondary

* Evaluate the trend of severity of radiation esophagitis-related pain during combined chemotherapy and radiation therapy for lung cancer using weekly measurements of the NRPS.
* Evaluate the adverse events associated with Manuka honey, as measured by CTCAE, v. 4.
* Evaluate the severity of radiation esophagitis (grade 3-4, CTCAE, v. 4).
* Assess weight loss (percent weight change from baseline to 4 weeks).
* Assess quality of life (QOL) and pain, as measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-30) global QOL score and pain symptom subscale.
* Assess patient-reported dysphagia via a daily patient log.
* Assess nutritional status, as measured by the mean change in serum prealbumin levels from baseline to 4 weeks.
* Assess opioid use by collecting the patient's narcotic use in the previous 24-hour period at each weekly evaluation.
* Evaluate patient-reported adverse events associated with Manuka honey using the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).

OUTLINE: This is a multicenter study. Patients are stratified according to the percentage of esophagus in the radiation field (V60 < 30% vs V60 ≥ 30%). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive standard supportive care for esophagitis-related pain as needed during chemoradiotherapy.
* Arm II: Patients swallow liquid Manuka honey slowly over 3-5 minutes. Patients must refrain from eating and drinking for 1 hour after administration. Treatment continues 4 times per day during chemoradiotherapy.
* Arm III: Patients place Manuka honey lozenges in their mouth one at a time and swallow the honey as it dissolves (no chewing or swallowing it whole). Patients must refrain from eating and drinking for 1 hour after administration. Treatment continues 4 times per day during chemoradiotherapy.

Patients complete quality of life, pain swallowing diary, and pain assessments (Numerical Rating Pain Scale, EORTC QLQ-30 and Pain Subscale, and PRO-CTCAE) periodically during study treatment.

Patients are followed up at 12 weeks from the start of study treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients being treated with combination chemotherapy (definitive or adjuvant) and radiation therapy once daily for small cell or non-small cell lung cancer (primary population for the trial)

  * Patients can receive chemoradiotherapy while on a Radiation Therapy Oncology Group (RTOG) lung trial or while not being on a clinical trial
  * No patients receiving chemoradiotherapy while enrolled on a single institution trial or trials coordinated by other cooperative groups
* No patients with metastatic disease
* At least 5 cm of the esophagus must be in the 60 Gy isodose volume in 1.6 to 2.0 Gy fractions

PATIENT CHARACTERISTICS:

* Age 18 and up
* Able to swallow thick liquids prior to treatment
* Able to speak English or Spanish in order to complete required forms (verbal completion is adequate)
* No patients with poorly controlled diabetes
* No known hypersensitivity to honey

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No patients who have received prior chemotherapy or radiation therapy
* No patients receiving more than once daily treatments
* Therapeutic use of honey other than the Manuka honey provided for this trial is not allowed while patients are on study
* Patients must also avoid honey-flavored medical products and/or sugary, viscous substances
* Amifostine is not permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence B. Berk, MD, PhD, Principal Investigator — Tampa General Hospital, University of South Florida
Locations (59):
- United States (59):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Cape Cod Hospital, Hyannis, Massachusetts
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - Payson Center for Cancer Care at Concord Hospital, Concord, New Hampshire
  - Seacoast Cancer Center at Wentworth - Douglass Hospital, Dover, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Trinity CancerCare Center, Minot, North Dakota
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - St. Joseph Cancer Center, Bellingham, Washington
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Supportive Care: Standard supportive care for esophagitis-related pain as needed during concurrent chemotherapy and radiation treatment.
- Liquid Manuka Honey: Manuka honey in liquid form during concurrent chemotherapy and radiation treatment.
- Lozenge Manuka Honey: Manuka honey in lozenge form during concurrent chemotherapy and radiation treatment.
Period: Overall Study
Arm/Group | Supportive Care | Liquid Manuka Honey | Lozenge Manuka Honey
Started | 53 | 54 | 56
Completed | 53 (Randomized eligible patients who received protocol treatment.) | 53 (Randomized eligible patients who received protocol treatment.) | 54 (Randomized eligible patients who received protocol treatment.)
Not Completed | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Supportive Care | Liquid Manuka Honey | Lozenge Manuka Honey | Total
Number analyzed (Participants) | 53 | 53 | 54 | 160
Age, Continuous [Median (Full Range); unit: years] | 65 [45 to 85] | 66 [37 to 83] | 65 [47 to 83] | 65 [37 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 23 | 74
  Male | 26 | 29 | 31 | 86

OUTCOME MEASURES:

1. Primary Outcome: Change in Radiation Esophagitis-related Pain at 4 Weeks as Measured by the Numerical Rating Pain Scale for Pain on Swallowing (NRPS)
Description: Esophagitis-related pain was measured using patient-reported pain on swallowing as assessed by the Numerical Rating Pain Scale (NRPS), an 11-point scale (0-10) in which 0 indicates no pain and 10 indicates the worst pain imaginable. Generally, scores of 1-4 indicate mild pain, scores of 5-6 indicate moderate pain, and scores of 7-10 indicate severe pain. Change was calculated by subtracting the baseline value from the 4-week value. The experimental arms (honey) were compared to the standard arm (supportive care).
Time Frame: Baseline and 4 weeks from the start of treatment
Population: Randomized eligible patients with NRPS score at both baseline and 4 weeks.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care | Liquid Manuka Honey | Lozenge Manuka Honey
Number analyzed (Participants) | 40 | 41 | 38
units on a scale | 1 [0 to 4] | 1 [0 to 4] | 1 [0 to 4]
Statistical Analysis 1: Comparison: Supportive Care vs Liquid Manuka Honey; Null hypothesis: Manuka honey in liquid form is/not effective at reducing esophagitis-related pain, measured by mean change score from 0 to 4 weeks. A 2-sample t-test for difference of means with alpha 0.05 after adjusting for multiple comparisons (1-sided with overall alpha 0.1 before the Bonferroni adjustment) and 80% statistical power for each hypothesis test requires 45 patients per arm to detect >= 15% relative reduction (absolute difference of mean change score of 3.1; effect size=0.53); Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney) — Due to the skewed nature of the data, median was reported instead of mean; Each arm had less than the designed sample size. Therefore the statistical power was reduced (76% instead of 80%)
Statistical Analysis 2: Comparison: Supportive Care vs Lozenge Manuka Honey; Null hypothesis: Manuka honey in lozenge form is/not effective at reducing esophagitis-related pain, measured by mean change score from 0 to 4 weeks. A 2-sample t-test for difference of means with alpha 0.05 after adjusting for multiple comparisons (1-sided with overall alpha 0.1 before the Bonferroni adjustment) and 80% statistical power for each hypothesis test requires 45 patients per arm to detect >= 15% relative reduction (absolute difference of mean change score of 3.1; effect size=0.53); Test type: Superiority or Other; p = 0.93, Wilcoxon (Mann-Whitney) — Due to the skewed nature of the data, median was reported instead of mean; Each arm had less than the designed sample size. Therefore the statistical power was reduced (76% instead of 80%)

2. Secondary Outcome: Radiation Esophagitis-related Pain During Treatment as Measured During Treatment and 12 Weeks by the Numerical Rating Pain Scale (NRPS)
Description: Esophagitis-related pain was measured using patient-reported pain on swallowing as assessed by the Numerical Rating Pain Scale (NRPS), an 11-point scale (0-10) in which 0 indicates no pain and 10 indicates the worst pain imaginable. Generally, scores of 1-4 indicate mild pain, scores of 5-6 indicate moderate pain, and scores of 7-10 indicate severe pain. Change was calculated by subtracting the baseline value from values at the later time points. The experimental arms (honey) were compared to the standard arm (supportive care).
Time Frame: Baseline, weekly during treatment, and 12 weeks from the start of treatment
Population: Eligible patients who started protocol treatment with at least 1 NRPS score completed across all time points
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care | Liquid Manuka Honey | Lozenge Manuka Honey
Number analyzed (Participants) | 49 | 50 | 51
units on a scale
  Baseline: number analyzed (Participants) | 48 | 50 | 51
  Baseline | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Week 1: number analyzed (Participants) | 41 | 42 | 38
  Week 1 | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 0]
  Week 2: number analyzed (Participants) | 41 | 42 | 38
  Week 2 | 0 [0 to 2] | 0 [0 to 1] | 0 [0 to 3]
  Week 3: number analyzed (Participants) | 42 | 42 | 39
  Week 3 | 0 [0 to 4] | 1 [0 to 4] | 1 [0 to 3]
  4 weeks: number analyzed (Participants) | 43 | 43 | 39
  4 weeks | 1 [0 to 4] | 1 [0 to 4] | 2 [0 to 5]
  Week 5: number analyzed (Participants) | 36 | 40 | 37
  Week 5 | 2.5 [0 to 4.5] | 2 [0 to 5] | 3 [0 to 6]
  End of RT: number analyzed (Participants) | 37 | 40 | 38
  End of RT | 3 [0 to 5.5] | 3 [0 to 6] | 4 [0 to 6]
  Week 12: number analyzed (Participants) | 37 | 36 | 40
  Week 12 | 0 [0 to 2] | 0 [0 to 2.5] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with NRPS score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Treatment (Liquid Honey vs. Supportive Care) is reported here; Test type: Superiority or Other; p = 0.87, Mixed Models Analysis; Explanatory variables are reported separately
Statistical Analysis 2: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with NRPS score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Treatment (Lozenge Honey vs. Supportive Care) is reported here; Test type: Superiority; p = 0.46, Mixed Models Analysis; Each explanatory variable is reported separately
Statistical Analysis 3: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with NRPS score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Percentage of esophagus is reported here; Test type: Superiority; p = 0.0023, Mixed Models Analysis; Each explanatory variable is reported separately
Statistical Analysis 4: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with NRPS score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Opioid use is reported here; Test type: Superiority; p = 0.0025, Mixed Models Analysis; Each explanatory variable is reported separately
Statistical Analysis 5: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with NRPS score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Time is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Each explanatory variable is reported separately

3. Secondary Outcome: Dysphagia Via Daily Patient Log
Description: Dysphagia, as reported by the patient, was measured by the patient swallowing diary. Swallowing score has increasing severity 1-5, where 1 = "none" and 5 = "cannot swallow liquids".
Time Frame: Weekly during treatment and 12 weeks from the start of treatment
Population: Randomized eligible patients who received protocol treatment with at least one dysphagia score completed across all time points.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care | Liquid Manuka Honey | Lozenge Manuka Honey
Number analyzed (Participants) | 46 | 50 | 59
units on a scale
  Baseline: number analyzed (Participants) | 46 | 50 | 49
  Baseline | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Week 1: number analyzed (Participants) | 34 | 37 | 32
  Week 1 | 1 [1 to 1.14] | 1 [1 to 1] | 1 [1 to 1.29]
  Week 2: number analyzed (Participants) | 34 | 41 | 34
  Week 2 | 1 [1 to 1.57] | 1 [1 to 1.43] | 1.07 [1 to 2]
  Week 3: number analyzed (Participants) | 34 | 39 | 33
  Week 3 | 1.36 [1 to 2.43] | 2 [1 to 2.14] | 1.86 [1 to 2.86]
  Week 4: number analyzed (Participants) | 33 | 37 | 32
  Week 4 | 1.86 [1 to 2.86] | 2 [1 to 2.57] | 2.07 [1.15 to 3]
  Week 5: number analyzed (Participants) | 32 | 37 | 30
  Week 5 | 2.5 [1.07 to 3] | 2 [1 to 3] | 2.71 [2 to 3]
  End of RT: number analyzed (Participants) | 30 | 33 | 26
  End of RT | 2 [1 to 3] | 2.86 [1.71 to 3] | 3 [2.86 to 3.71]
  Week 12: number analyzed (Participants) | 36 | 38 | 36
  Week 12 | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with dysphagia score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. Treatment (Liquid Honey vs. Supportive Care) is reported here; Test type: Superiority or Other; p = 0.70, Mixed Models Analysis; Explanatory variables are reported separately
Statistical Analysis 2: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with dysphagia score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Treatment (Lozenge Honey vs. Supportive Care) is reported here; Test type: Superiority or Other; p = 0.71, Mixed Models Analysis; Explanatory variables are reported separately
Statistical Analysis 3: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with dysphagia score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Percentage of esophagus is reported here; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Each explanatory variable is reported separately
Statistical Analysis 4: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with dysphagia score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Opioid use is reported here; Test type: Superiority; p = 0.0051, Mixed Models Analysis; Each explanatory variable is reported separately
Statistical Analysis 5: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with dysphagia score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Time is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately

4. Secondary Outcome: Quality of Life and Pain, as Measured by the EORTC QLQ-30 Global QOL Score and Pain Symptom Subscale at 4 and 12 Weeks
Description: The pain symptom subscale (2 items) evaluated pain and the global score (30 items) evaluated quality of life. Each ranges from 0-100 with lower scores indicating lesser burden and improved symptoms or quality of life.
Time Frame: Baseline, 4 and 12 weeks from the start of treatment
Population: Randomized eligible patients who received protocol treatment with at least 1 EORTC score completed across all time points.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care | Liquid Manuka Honey | Lozenge Manuka Honey
Number analyzed (Participants) | 48 | 50 | 52
units on a scale
  Baseline - Global health status | 66.67 [54.17 to 83.33] | 66.67 [50.00 to 83.33] | 66.67 [50.00 to 83.33]
  Baseline - Pain | 16.67 [0 to 41.67] | 16.67 [0 to 33.33] | 16.67 [0 to 50.00]
  Week 4 - Global health status: number analyzed (Participants) | 38 | 40 | 43
  Week 4 - Global health status | 66.67 [50.00 to 75.00] | 62.50 [45.83 to 75.00] | 66.67 [50.00 to 75.00]
  Week 4 - Pain: number analyzed (Participants) | 38 | 40 | 43
  Week 4 - Pain | 25.00 [0.00 to 33.33] | 16.67 [0.00 to 50.00] | 33.33 [0.00 to 50.00]
  Week 12 - Global health status: number analyzed (Participants) | 37 | 38 | 39
  Week 12 - Global health status | 66.67 [50.00 to 83.33] | 58.33 [41.67 to 83.33] | 66.67 [41.67 to 83.33]
  Week 12 - Pain: number analyzed (Participants) | 37 | 38 | 39
  Week 12 - Pain | 0.00 [0.00 to 33.33] | 16.67 [0.00 to 33.33] | 16.67 [0.00 to 33.33]
Statistical Analysis 1: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with EORTC global health status (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Treatment (Liquid Honey vs. Supportive Care) is reported here; Test type: Superiority or Other; p = 0.086, Mixed Models Analysis; Explanatory variables are reported separately
Statistical Analysis 2: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with EORTC global health status (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Treatment (Lozenge Honey vs. Supportive Care) is reported here; Test type: Superiority or Other; p = 0.20, Mixed Models Analysis; Each explanatory variable is reported separately
Statistical Analysis 3: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with EORTC global health status (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Percentage of esophagus is reported here; Test type: Superiority; p = 0.44, Mixed Models Analysis; Each explanatory variable is reported separately
Statistical Analysis 4: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with EORTC global health status (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Opioid use is reported here; Test type: Superiority; p = 0.0066, Mixed Models Analysis; Each explanatory variable is reported separately
Statistical Analysis 5: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with EORTC global health status (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Time is reported here; Test type: Superiority; p = 0.36, Mixed Models Analysis; Each explanatory variable is reported separately
Statistical Analysis 6: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with EORTC pain score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Treatment (Liquid Honey vs. Supportive Care) is reported here; Test type: Superiority or Other; p = 0.94, Mixed Models Analysis; Explanatory variables are reported separately
Statistical Analysis 7: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with EORTC pain score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Treatment (Lozenge Honey vs. Supportive Care) is reported here; Test type: Superiority or Other; p = 0.58, Mixed Models Analysis; Each explanatory variable is reported separately
Statistical Analysis 8: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with EORTC pain score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Percentage of esophagus is reported here; Test type: Superiority; p = 0.28, Mixed Models Analysis; Each explanatory variable is reported separately
Statistical Analysis 9: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with EORTC pain score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Opioid use is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each exploratory variable is reported separately
Statistical Analysis 10: Comparison: Supportive Care vs Liquid Manuka Honey vs Lozenge Manuka Honey; A linear fixed effects model using maximum likelihood estimation was run with EORTC pain score (baseline, weekly during treatment and 12 weeks from the end of treatment) as the outcome of interest. Percentage of esophagus (V60>=30% as reference level), opioid use ("yes" as reference level), time, and treatment arm were factors in the model. The results for each explanatory variable are reported separately. Time is reported here; Test type: Superiority; p = 0.28, Mixed Models Analysis; Each explanatory variable is reported separately

5. Secondary Outcome: Percentage of Participants With Radiation Esophagitis Grade 3-4 (CTCAE v. 4)
Description: Adverse events are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. For esophagitis specifically, Grade 3 criteria includes severely altered eating/swallowing, tube feeding, total parenteral nutrition (TPN) or hospitalization indicated. Grade 4 criteria include life-threatening consequences, urgent operative intervention indicated.
Time Frame: Up to 12 weeks from the start of treatment
Population: Randomized eligible patients who started protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supportive Care | Liquid Manuka Honey | Lozenge Manuka Honey
Number analyzed (Participants) | 48 | 50 | 50
percentage of participants | 12.5 [3.1 to 21.9] | 2.0 [0.0 to 5.9] | 6.0 [0.0 to 12.6]
Statistical Analysis 1: Comparison: Supportive Care vs Liquid Manuka Honey; Test type: Superiority or Other; p = 0.06, Fisher Exact — Significance level = 0.05
Statistical Analysis 2: Comparison: Supportive Care vs Lozenge Manuka Honey; Test type: Superiority or Other; p = 0.31, Fisher Exact — Significance level = 0.05

6. Secondary Outcome: Percent Change in Weight From Baseline to 4 Weeks
Time Frame: Baseline and 4 weeks from the start of treatment
Population: Randomized eligible patients with weight at both baseline and 4 weeks.
Measure: Mean (95% Confidence Interval); unit: percentage of baseline value
Arm/Group | Supportive Care | Liquid Manuka Honey | Lozenge Manuka Honey
Number analyzed (Participants) | 50 | 51 | 51
percentage of baseline value | -2.22 [-7.26 to 14.79] | -0.62 [-1.57 to 2.83] | -2.64 [-4.53 to 5.64]
Statistical Analysis 1: Comparison: Supportive Care vs Liquid Manuka Honey; Test type: Superiority or Other; p = 0.53, t-test, 2 sided — significance level = 0.05
Statistical Analysis 2: Comparison: Supportive Care vs Lozenge Manuka Honey; Test type: Superiority or Other; p = 0.88, t-test, 2 sided — significance level = 0.05

7. Secondary Outcome: Nutritional Status (Change in Serum Prealbumin Levels From Baseline to 4 Weeks)
Time Frame: Baseline and 4 weeks from the start of treatment
Population: Randomized eligible patients with serum prealbumin at baseline and 4 weeks.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Supportive Care | Liquid Manuka Honey | Lozenge Manuka Honey
Number analyzed (Participants) | 50 | 51 | 51
mg/dl | -3.34 [-9.46 to 17.98] | 5.25 [-6.42 to 34.70] | 0.17 [-1.94 to 6.28]
Statistical Analysis 1: Comparison: Supportive Care vs Liquid Manuka Honey; Test type: Superiority or Other; p = 0.20, t-test, 2 sided
Statistical Analysis 2: Comparison: Supportive Care vs Lozenge Manuka Honey; Test type: Superiority or Other; p = 0.28, t-test, 2 sided

8. Secondary Outcome: Percentage of Patients Using Opioids
Description: The percentage of patients using opioid analgesics is reported. Use of opioid analgesics was assessed for a 24-hour period before completing the assessment. Patients with at least one reported administration of opioid analgesic were considered to have received opioid analgesics.
Time Frame: Baseline, 4 weeks, end of radiation treatment, and 12 weeks from the start of treatment
Population: Randomized eligible patients with opioid use information at at least one time point.
Measure: Number; unit: percentage of participants
Arm/Group | Supportive Care | Liquid Manuka Honey | Lozenge Manuka Honey
Number analyzed (Participants) | 53 | 53 | 54
percentage of participants
  Baseline | 13.2 | 9.4 | 13.0
  Week 4: number analyzed (Participants) | 46 | 49 | 48
  Week 4 | 37.0 | 14.3 | 29.2
  End of RT: number analyzed (Participants) | 43 | 47 | 44
  End of RT | 46.5 | 36.2 | 43.2
  Week 12: number analyzed (Participants) | 43 | 46 | 44
  Week 12 | 32.6 | 17.4 | 18.2

9. Secondary Outcome: Adverse Events Associated With Manuka Honey Using CTCAE v4.0
Description: Adverse events are graded using CTCAE v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: Until 12 weeks from the start of treatment
Population: Randomized eligible patients who started protocol treatment.
Measure: Number; unit: percentage of patients
Arm/Group | Supportive Care | Liquid Manuka Honey | Lozenge Manuka Honey
Number analyzed (Participants) | 48 | 50 | 50
percentage of patients
  Grade 1 | 6.3 | 16.0 | 12.0
  Grade 2 | 20.8 | 26.0 | 18.0
  Grade 3 | 10.4 | 8.0 | 8.0
  Grade 4 | 2.1 | 0.0 | 2.0
  Grade 5 | 0.0 | 0.0 | 0.0

10. Secondary Outcome: Patient Reported Difficulty in Swallowing Associated With Manuka Honey Using the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: Change from baseline to four weeks in patient-reported difficulty in swallowing via the PRO-CTCAE. PRO-CTCAE is an item bank consisting of individual items to assess adverse symptom events from the patient perspective. There are 78 symptoms included in the survey but the primary item of interest assesses difficulty swallowing. For each AE in the PRO-CTCAE, between 1 and 3 items are included to assess the frequency, severity, and/or interference with activities related to that AE. Frequency questions have responses ranging from never, which is scored as a 0, to almost constantly, which is scored as a 4. Severity questions have responses ranging from none, which is scored as a 0, to very severe, which is scored as a 4. Interference questions have responses ranging from not at all, which is scored as a 0, to very much, which is scored as a 4. Difficulty in swallowing only has a severity question.
Time Frame: Baseline and 4 weeks from the start of treatment
Population: Randomized eligible patients who started treatment with measure at both baseline and 4 weeks.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care | Liquid Manuka Honey | Lozenge Manuka Honey
Number analyzed (Participants) | 36 | 33 | 35
units on a scale | 1 [0 to 2] | 1 [0 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: Supportive Care vs Liquid Manuka Honey; Each experimental arm was compared to the control arm (i.e. 2 comparisons) using two-sample t-tests. Forty-five patients with data in each arm, provides 80% power to detect an effect size (in standard deviation units) of 0.60 and 90% power to detect an effect size of 0.69 using a two-sided T-test with a Bonferroni adjusted significance level of 0.05 for each comparison (overall alpha 0.10). Due to the lack of prior data on the PRO-CTCAE, moderate effect sizes were used; Test type: Superiority or Other; p = 0.39, Wilcoxon (Mann-Whitney); Because data was not normally distributed, this test was used instead of the t-test
Statistical Analysis 2: Comparison: Supportive Care vs Lozenge Manuka Honey; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.69, Wilcoxon (Mann-Whitney); Because data was not normally distributed, this test was used instead of the t-test

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Supportive Care | Liquid Manuka Honey | Lozenge Manuka Honey
Serious Adverse Events (participants affected / at risk) | 16/48 | 13/50 | 9/50
Other Adverse Events (participants affected / at risk) | 37/48 | 46/50 | 38/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Supportive Care (N=48) | Liquid Manuka Honey (N=50) | Lozenge Manuka Honey (N=50)
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 3
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 5 | 1 | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0
Infusion related reaction (General disorders) | 1 | 0 | 0
Lung infection (Infections and infestations) | 2 | 0 | 2
Sepsis (Infections and infestations) | 1 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 2 | 2
Platelet count decreased (Investigations) | 1 | 2 | 1
Weight loss (Investigations) | 0 | 1 | 0
White blood cell decreased (Investigations) | 1 | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nervous system disorders - Other (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Supportive Care (N=48) | Liquid Manuka Honey (N=50) | Lozenge Manuka Honey (N=50)
Anemia (Blood and lymphatic system disorders) | 15 | 20 | 13
Constipation (Gastrointestinal disorders) | 13 | 15 | 10
Diarrhea (Gastrointestinal disorders) | 9 | 11 | 3
Dry mouth (Gastrointestinal disorders) | 3 | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 10 | 6 | 2
Dysphagia (Gastrointestinal disorders) | 17 | 20 | 17
Esophageal pain (Gastrointestinal disorders) | 2 | 8 | 3
Esophagitis (Gastrointestinal disorders) | 19 | 18 | 13
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 5 | 3
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 3 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 2 | 5
Nausea (Gastrointestinal disorders) | 16 | 23 | 11
Vomiting (Gastrointestinal disorders) | 7 | 6 | 4
Fatigue (General disorders) | 28 | 28 | 22
Non-cardiac chest pain (General disorders) | 1 | 3 | 0
Pain (General disorders) | 3 | 6 | 4
Mucosal infection (Infections and infestations) | 0 | 3 | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 12 | 7 | 11
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 | 3 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 4
Alkaline phosphatase increased (Investigations) | 2 | 3 | 1
Creatinine increased (Investigations) | 2 | 5 | 3
Lymphocyte count decreased (Investigations) | 7 | 5 | 2
Neutrophil count decreased (Investigations) | 6 | 7 | 10
Platelet count decreased (Investigations) | 4 | 9 | 11
Weight loss (Investigations) | 4 | 8 | 3
White blood cell decreased (Investigations) | 8 | 13 | 8
Anorexia (Metabolism and nutrition disorders) | 10 | 17 | 5
Dehydration (Metabolism and nutrition disorders) | 6 | 8 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 7 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 5 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 5 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 3 | 3
Hyponatremia (Metabolism and nutrition disorders) | 4 | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1
Dizziness (Nervous system disorders) | 3 | 5 | 2
Dysgeusia (Nervous system disorders) | 6 | 8 | 4
Headache (Nervous system disorders) | 5 | 4 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 3 | 2
Anxiety (Psychiatric disorders) | 4 | 3 | 2
Depression (Psychiatric disorders) | 1 | 4 | 0
Insomnia (Psychiatric disorders) | 6 | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 22 | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 17 | 13
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 3 | 1
Hypotension (Vascular disorders) | 1 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.